CLINICAL TRIAL: NCT02045121
Title: A Multicentre Randomised Study Comparing Indwelling Pleural Catheter With Talc Pleurodesis in Patients With a Malignant Pleural Effusion
Brief Title: Multicentre Study Comparing Indwelling Pleural Catheter With Talc Pleurodesis for Malignant Pleural Effusion Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, A/Prof Lee Pyng, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSRG/0042/2013
Record Dates: First submitted 2014-01-09; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant

ARMS (2):
- Indwelling Pleural Catheter (Experimental): Day-case IPC insertion. Attendance d10 for drainage, stitch removal and education in catheter care.
  Interventions: Device: Indwelling Pleural Catheter
- Talc Pleurodesis (Active Comparator): Hospital admission for chest drain insertion and suction if needed, plus talc pleurodesis by slurry or poudrage if >75% of visceral and parietal pleura in direct contact on chest x-ray.
  Interventions: Procedure: Talc Pleurodesis

INTERVENTIONS:
Device: Indwelling Pleural Catheter
  Arms: Indwelling Pleural Catheter
Procedure: Talc Pleurodesis
  Arms: Talc Pleurodesis

SUMMARY:
Malignant pleural effusion (MPE) accounts for 50% of all pleural effusions and affects about 300,000 patients annually (UK and USA). Lung and breast cancers account for majority of malignant pleural effusions; 1 in 3 breast cancer, 1 in 4 lung cancer as well as > 90% of patients with mesothelioma develop pleural effusions. Breathlessness from MPE is disabling and impairs quality of life. Median survival ranges between 4-6 months. Although thoracentesis provides effective symptom relief, most effusions recur and pleurodesis is the standard of care. Pleurodesis can be performed via chest tube or applied during pleuroscopy, and talc is the most effective agent. For successful pleurodesis to occur the underlying lung must expand after fluid drainage and trapped lung due to metastatic disease occurs up to 30%. Symptomatic patients require hospitalization for these procedures which are likely to fail if trapped lungs are encountered, and pose significant burden to health services. Tunneled indwelling pleural catheter (IPC) is emerging as a viable alternative which provides access to the pleural space for fluid drainage when breathlessness arise. IPC can be performed at ambulatory setting without hospital admission. Case series have demonstrated long-term safety of IPC even in patients undergoing chemotherapy with acceptable complication rates. By keeping the pleural cavity free of fluid, IPC has led to spontaneous pleurodesis in 50% of patients, which allows its removal. Presently IPC is indicated for trapped lung or when talc pleurodesis has failed. A randomised comparative trial with talc pleurodesis is necessary to determine role of IPC as first-line therapy of MPE, if IPC leads to reduction in hospitalizations, adverse events and healthcare costs, and if it improves quality of life. The multicenter trial randomizes symptomatic patients 1:1 to IPC or talc pleurodesis, and endpoints include hospitalization days till death or end of study, adverse events, quality of life, and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic malignant pleural effusion requiring intervention

Exclusion Criteria:

* <18 years of age
* pregnant or lactating patients
* expected survival <3 months
* chylothorax
* previous attempted pleurodesis
* pleural infection
* leukocytopaenia (<1.0 x 10^9/L)
* uncorrectable bleeding diathesis
* inability to give informed consent or comply with the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Number of hospital days for all causes following intervention | Up to 1 year

SECONDARY OUTCOMES:
Number of hospital days computed for pleural effusion related cause | Up to 1 year
Number of adverse events | Up to 1 year
Breathlessness score | Up to 1 year
Self-reported quality of life scores | Up to 1 year
Health costs computation | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pyng Lee, MBBS, MRCP, MMED, FAMS, FCCP, Principal Investigator — National University of Singapore
Locations (1):
- Division of Respiratory and Critical Care Medicine, National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Davies HE, Lee YCG. Pleurodesis. In: Light RW, Lee YCG, eds. Textbook of Pleural Diseases. 2nd ed. London, U.K.: Arnold Press; 2008:569-82.
- [Background] Mishra E, Davies HE, Lee YCG. Malignant pleural disease in primary lung cancer. In: Spiro SG, Janes SM, Huber RM, eds. Thoracic Malignancies. 3rd ed ed. Sheffield, U.K.: European Respiratory Society Journals Ltd; 2009:318-35.
- [Background] Lee YC, Wilkosz S. Malignant pleural effusions: fixing the leaky faucet. Am J Respir Crit Care Med. 2008 Jul 1;178(1):3-5. doi: 10.1164/rccm.200804-616ED. No abstract available. PMID 18565960
- [Background] West SD, Lee YC. Management of malignant pleural mesothelioma. Clin Chest Med. 2006 Jun;27(2):335-54. doi: 10.1016/j.ccm.2006.01.004. PMID 16716822
- [Background] Burrows CM, Mathews WC, Colt HG. Predicting survival in patients with recurrent symptomatic malignant pleural effusions: an assessment of the prognostic values of physiologic, morphologic, and quality of life measures of extent of disease. Chest. 2000 Jan;117(1):73-8. doi: 10.1378/chest.117.1.73. PMID 10631202
- [Background] Heffner JE, Nietert PJ, Barbieri C. Pleural fluid pH as a predictor of survival for patients with malignant pleural effusions. Chest. 2000 Jan;117(1):79-86. doi: 10.1378/chest.117.1.79. PMID 10631203
- [Background] Robinson BW, Musk AW, Lake RA. Malignant mesothelioma. Lancet. 2005 Jul 30-Aug 5;366(9483):397-408. doi: 10.1016/S0140-6736(05)67025-0. PMID 16054941
- [Background] Dresler CM, Olak J, Herndon JE 2nd, Richards WG, Scalzetti E, Fleishman SB, Kernstine KH, Demmy T, Jablons DM, Kohman L, Daniel TM, Haasler GB, Sugarbaker DJ; Cooperative Groups Cancer and Leukemia Group B; Eastern Cooperative Oncology Group; North Central Cooperative Oncology Group; Radiation Therapy Oncology Group. Phase III intergroup study of talc poudrage vs talc slurry sclerosis for malignant pleural effusion. Chest. 2005 Mar;127(3):909-15. doi: 10.1378/chest.127.3.909. PMID 15764775
- [Background] Davies HE, Lee YC, Davies RJ. Pleurodesis for malignant pleural effusion: talc, toxicity and where next? Thorax. 2008 Jul;63(7):572-4. doi: 10.1136/thx.2007.092940. No abstract available. PMID 18587029
- [Background] Lee YC, Fysh ET. Indwelling pleural catheter: changing the paradigm of malignant effusion management. J Thorac Oncol. 2011 Apr;6(4):655-7. doi: 10.1097/JTO.0b013e3182114aa0. No abstract available. PMID 21623256
- [Background] van den Toorn LM, Schaap E, Surmont VF, Pouw EM, van der Rijt KC, van Klaveren RJ. Management of recurrent malignant pleural effusions with a chronic indwelling pleural catheter. Lung Cancer. 2005 Oct;50(1):123-7. doi: 10.1016/j.lungcan.2005.05.016. PMID 15998551
- [Background] Tremblay A, Mason C, Michaud G. Use of tunnelled catheters for malignant pleural effusions in patients fit for pleurodesis. Eur Respir J. 2007 Oct;30(4):759-62. doi: 10.1183/09031936.00164706. Epub 2007 Jun 13. PMID 17567670
- [Background] Putnam JB Jr, Walsh GL, Swisher SG, Roth JA, Suell DM, Vaporciyan AA, Smythe WR, Merriman KW, DeFord LL. Outpatient management of malignant pleural effusion by a chronic indwelling pleural catheter. Ann Thorac Surg. 2000 Feb;69(2):369-75. doi: 10.1016/s0003-4975(99)01482-4. PMID 10735665
- [Background] Putnam JB Jr, Light RW, Rodriguez RM, Ponn R, Olak J, Pollak JS, Lee RB, Payne DK, Graeber G, Kovitz KL. A randomized comparison of indwelling pleural catheter and doxycycline pleurodesis in the management of malignant pleural effusions. Cancer. 1999 Nov 15;86(10):1992-9. PMID 10570423
- [Background] Suzuki K, Servais EL, Rizk NP, Solomon SB, Sima CS, Park BJ, Kachala SS, Zlobinsky M, Rusch VW, Adusumilli PS. Palliation and pleurodesis in malignant pleural effusion: the role for tunneled pleural catheters. J Thorac Oncol. 2011 Apr;6(4):762-7. doi: 10.1097/JTO.0b013e31820d614f. PMID 21325982
- [Background] Van Meter ME, McKee KY, Kohlwes RJ. Efficacy and safety of tunneled pleural catheters in adults with malignant pleural effusions: a systematic review. J Gen Intern Med. 2011 Jan;26(1):70-6. doi: 10.1007/s11606-010-1472-0. Epub 2010 Aug 10. PMID 20697963
- [Background] Morel A, Mishra E, Medley L, Rahman NM, Wrightson J, Talbot D, Davies RJ. Chemotherapy should not be withheld from patients with an indwelling pleural catheter for malignant pleural effusion. Thorax. 2011 May;66(5):448-9. doi: 10.1136/thx.2009.133504. Epub 2010 Sep 29. No abstract available. PMID 20880866
- [Background] Janes SM, Rahman NM, Davies RJ, Lee YC. Catheter-tract metastases associated with chronic indwelling pleural catheters. Chest. 2007 Apr;131(4):1232-4. doi: 10.1378/chest.06-2353. PMID 17426232
- [Derived] Fysh ET, Thomas R, Read CA, Kwan BC, Yap E, Horwood FC, Lee P, Piccolo F, Shrestha R, Garske LA, Lam DC, Rosenstengel A, Bint M, Murray K, Smith NA, Lee YC. Protocol of the Australasian Malignant Pleural Effusion (AMPLE) trial: a multicentre randomised study comparing indwelling pleural catheter versus talc pleurodesis. BMJ Open. 2014 Nov 6;4(11):e006757. doi: 10.1136/bmjopen-2014-006757. PMID 25377015